CLINICAL TRIAL: NCT03729804
Title: A Randomized, Open-label Phase 3 Study of Carfilzomib, Lenalidomide, and Dexamethasone Versus Bortezomib, Lenalidomide and Dexamethasone (KRd vs. VRd) in Patients With Newly Diagnosed Multiple Myeloma (COBRA)
Brief Title: Carfilzomib, Lenalidomide, and Dexamethasone Versus Bortezomib, Lenalidomide and Dexamethasone (KRd vs. VRd) in Patients With Newly Diagnosed Multiple Myeloma (COBRA)
Acronym: (COBRA)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-1243
Record Dates: First submitted 2018-10-12; First posted 2018-11-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KRD Arm (Experimental): Patients assigned to this group will receive a combination of carfilzomib, lenalidomide, and dexamethasone in 28 day cycles. Doses will vary
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- VRD Arm (Experimental): Patients assigned to this group will receive a combination of Bortezomib, lenalidomide and dexamethasone in 21-day cycles. Doses will vary
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be given by IV on Days 1, 2, 15 and 16 of each cycle during cycles 1-8.
  Carfilzomib will be given by IV on days 1, 2, 15 and 16 of each cycle during cycles 9-24.
  Other Names: Kyprolis
  Arms: KRD Arm
Drug: Lenalidomide — Lenalidomide will be taken by mouth once a day for days 1-21 of each cycle during cycles 1-8.
  Lenalidomide will be taken by mouth once a day for days 1-21 of each cycle for cycles 9-24.
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — Dexamethasone will be taken by mouth on days 1, 8, 15 and 22 of each cycle during cycles 1-8.
  Dexamethasone will be taken by mouth on Days 1, 8, 15 and 22 of each cycle during cycles 9-24.
Drug: Bortezomib — Bortezomib will be give by IV on days 1, 4, 8 and 11 of each cycle during cycles 1-8.
  Other Names: Velcade; PS-341
  Arms: VRD Arm

SUMMARY:
This is a randomized multicenter study that will compare two treatment regimens (Kyprolis, Revlimid, dexamethasone -KRD vs. Velcade, Revlimid, dexamethasone -VRD) for patients with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, previously untreated myeloma requiring systemic chemotherapy per International Myeloma Working Group criteria:

   • Patients must have received no prior chemotherapy for this disease; patients must have received no prior radiotherapy to a large area of the pelvis (more than half of the pelvis); prior steroid treatment is allowed provided treatment was not more than 2 weeks in duration and less than or equal to 160 mg dexamethasone; patients must not have received any prior treatment with bortezomib or lenalidomide
2. Both transplant and non-transplant candidates are eligible. Transplant candidates must agree to defer transplant at time of consent.
3. Diagnosis of symptomatic multiple myeloma as per current International Myeloma Working Group uniform criteria prior to initial treatment
4. Monoclonal plasma cells in the BM 10% or presence of a biopsy-proven plasmacytoma
5. Measurable disease, prior to initial treatment as indicated by one or more of the following:

   * Serum M-protein greater than or equal to 1 g/dL
   * Urine M-protein greater than or equal to 200 mg/24 hours
   * If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable
6. Bone marrow specimen will be required at study entry; available DNA sample from pre-induction BM will be used for calibration step for Minimal Residual Disease evaluation by gene sequencing.
7. Males and females 18 years of age or older.
8. Eastern Cooperative Oncology Group performance status of 0-1
9. Adequate hepatic function, with bilirubin less than or equal to 1.5 x ULN and aspirate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
10. ANC greater than or equal to 1.0 x 109/L, hemoglobin greater than or equal to 8 g/dL, platelet count greater than or equal to 75 x 109/L.
11. Calculated creatinine clearance (by Cockroft-Gault) greater than or equal to 50 mL/min or serum creatinine below 2 g/dL
12. FCBP must have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to initiating lenalidomide. The first pregnancy test must be performed within 10-14 days before and the second pregnancy test must be performed within 24 hours before lenalidomide is prescribed for Cycle 1 (prescriptions must be filled within 7 days).
13. FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study; and 3) for at least 30 days after discontinuation from the study.
14. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 90 days following discontinuation from the study even if he has undergone a successful vasectomy.
15. All study participants in the US must be consented to and registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS®.
16. Subjects must comply with pregnancy prevention and counseling
17. Voluntary written informed consent.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study.

1. Frail non-transplant candidates, defined as in Palumbo et al, Blood 2015
2. Non-secretory or hyposecretory multiple myeloma, prior to initial treatment defined as less than 1.0 g/dL M-protein in serum, less than 200 mg/24 hr urine M-protein
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
4. Amyloidosis
5. Plasma cell leukemia
6. Waldenström's macroglobulinemia or IgM myeloma
7. Radiotherapy to multiple sites or immunotherapy within 4 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
8. Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater
9. Potential subjects with evidence of progressive disease as per IMWG criteria
10. Patients not able to tolerate daratumumab, carfilzomib, lenalidomide or dexamethasone
11. Peripheral neuropathy greater than or equal to Grade 2 at screening
12. Diarrhea greater than Grade 1 in the absence of antidiarrheals
13. CNS involvement
14. Patients who cannot undergo or unwilling to take thromoprophylaxis
15. Uncontrolled or symptomatic angina, arrhythmia, hypertension, CHF, EF less than 40%, within 6 months prior to first dose
16. Pregnant or lactating females
17. Major surgery within 3 weeks prior to first dose.
18. Myocardial infarction within 6 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
19. Prior or concurrent pulmonary embolism
20. Known moderate or severe persistent asthma or known chronic obstructive pulmonary disease (COPD)
21. Rate-corrected QT interval of electrocardiograph (QTc) greater than 470 msec on a 12-lead ECG during screening
22. Uncontrolled diabetes
23. Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
24. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
25. Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer less than Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
26. Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with progression free survival with the group taking KRd versus VRd after randomization | 5 years

SECONDARY OUTCOMES:
The rate of MRD-negative (minimal residual disease) at indicated time points of study after randomization | 5 years
The combination of drugs (KRd vs VRd) with the best response using minimal residual disease analysis across entire treatment in high risk and low risk patients | 5 years
The combination of drugs (KRd vs VRd) safety and tolerability based on patients response | 5 years
  The safety and tolerability of lenalidomide and carfilzomib will be evaluated by means of drug related Adverse Events reports.
Evaluate the correlation between treatment outcome using KRd or VRd and pre-treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided